CLINICAL TRIAL: NCT05368350
Title: Treating Primary Progressive Aphasia and Apraxia of Speech With High Definition Transcranial Direct Current Stimulation (HDtDCS-PPA/PAOS)
Brief Title: Treating Primary Progressive Aphasia and Apraxia of Speech Using Non-invasive Brain Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, John Hart, Jr., Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTD IRB: 24-595
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Primary Progressive Aphasia; Apraxia of Speech
MeSH Terms: conditions — Aphasia, Primary Progressive; Apraxias

STUDY DESIGN:
Masking Description: Study participants will be assigned to either Pre-SMA or LIFG arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Pre-SMA tDCS treatment (Experimental): This open-label treatment will examine improvement of speech output, verbal fluency, and other cognitive deficits associated with primary progressive aphasia (PPA) and progressive apraxia of speech (PAOS), by utilizing 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to pre-supplementary motor area for 20 minutes over 10 sessions. There will be baseline testing, and follow up testing immediately after and 8 weeks after completion of treatment.
  Interventions: Device: high-definition transcranial direct current stimulation (HD-tDCS)
- Active LIFG tDCS treatment (Experimental): This open-label treatment will examine improvement of speech output, verbal fluency, and other cognitive deficits associated with primary progressive aphasia (PPA) and progressive apraxia of speech (PAOS), by utilizing 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to left inferior frontal gyrus for 20 minutes over 10 sessions. There will be baseline testing, and follow up testing immediately after and 8 weeks after completion of treatment.
  Interventions: Device: high-definition transcranial direct current stimulation (HD-tDCS)

INTERVENTIONS:
Device: high-definition transcranial direct current stimulation (HD-tDCS) — Other Names:
  tDCS
  1 milliamp tDCS High definition tDCS High definition transcranial direct current stimulator, Neuroelectrics Starstim tES, SN E20200930-10 Transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. Stimulation will consist of 1 milliamp stimulation, with (1) Pre-SMA stimulation arm -- anodal stimulation delivered at electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns or (2) LIFG stimulation arm -- at electrode F7 (International 10/10 System for electroencephalography electrode placement) and electrodes T7, FP1, AF3, and FC5 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, then remain at 1 milliamp of stimulation over 20 minutes, and finally ramping down at to 0 milliamps over 60 seconds.

SUMMARY:
The purpose of the study is to test whether low level electric stimulation, called transcranial Direct Current Stimulation (tDCS), on the part of the brain (i.e., pre-supplementary motor area and left inferior frontal gyrus) thought to aid in memory will improve speech and language difficulties in patients with primary progressive aphasia (PPA) and progressive apraxia of speech (PAOS). The primary outcome measures are neuropsychological assessments of speech and language functions, and the secondary measures are neuropsychological assessments of other cognitive abilities and electroencephalography (EEG) measures.

DETAILED DESCRIPTION:
This pilot study has one treatment arm with open-label treatment and will examine improvement of speech output, verbal fluency, and other cognitive deficits associated with primary progressive aphasia (PPA) and progressive apraxia of speech (PAOS), by utilizing 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to pre-supplementary motor area or left inferior frontal gyrus for 20 minutes over 10 sessions. There will be baseline testing, and follow up testing immediately after and 8 weeks after completion of treatment.

All patients with a clinical diagnosis of PPA or PAOS will be assigned to either one of the two open-label arms to receive active tDCS. Primary outcome speech and language measures, secondary neuropsychological and electroencephalography (EEG) measures, and pre-screening assessments for study medical history and contraindications for treatment will be collected prior to the treatment (i.e., baseline).

Primary outcome speech and language functions measures and secondary neuropsychological and electroencephalography (EEG) measures will be collected after treatment session 10 and following treatment competition (i.e., 8-week).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age
* A formal diagnosis of primary progressive aphasia (nonfluent/agrammatic, semantic, logopenic variants or mixed) and/or progressive apraxia of speech
* Capable of understanding and signing an informed consent. Medical information/history, as well as mental status exam and diagnosis provided by referring physician will determine whether or not a caregiver is required to be involved during this process.

Exclusion Criteria:

* Has an implanted device, such as a pacemaker, metallic cranial implant, or a neurostimulator
* Skull defects
* Pregnant
* A significant history of arrhythmia or epileptic seizures.
* Not a native English speaker
* Currently receiving speech-language intervention
* Unable to communicated verbally

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-04-16 (Estimated); Study Completion 2026-04-16 (Estimated)

PRIMARY OUTCOMES:
The Controlled Oral Word Association Test | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on the Control Word Association Test
  Benton, L.A., Hamsher, K., & Sivan, A.B., (1994). Multilingual aphasia examination. Iowa City: AJA Associates.
Category Fluency | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on Category Fluency
  Benton, L.A., Hamsher, K., & Sivan, A.B., (1994). Multilingual aphasia examination. Iowa City: AJA Associates.
The Boston Naming Test | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on The Boston Naming Test (accuracy and speech latency)
  Kaplan, E., Goodglass, H., & Weintraub, S., (1983). Boston Naming Test (2nd ed.). Lea & Febiger: Philadelphia.
Spontaneous speech (content and fluency) of the Western Aphasia Battery-Revised | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on Spontaneous speech (content and fluency) of the Western Aphasia Battery-Revised
  Kertesz, Andrew. ( 1982). The Western aphasia battery. New York :Grune & Stratton.
The Apraxia battery for Adults - 2 (ABA - 2) | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on characteristics of articulation of the the Apraxia battery for Adults - 2
  Dabul, B. L. (2000). Apraxia Battery for Adults (ABA-2) (2nd edn). Austin, TX: ProEd.

SECONDARY OUTCOMES:
The Trail Making Test (Part A & B) | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on The Trail Making Test (Part A & B)
  Reitan, R.M., (1958). Validity of the Trail Making Test as an indicator of organic brain damage. Percept. Motor Skill., 8, 271-276.
The Digit Span Forward & Backward | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on The Digit Span Forward & Backward
  Wechsler, D., (2008). Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio, TX: NCS Pearson.
The Digit Symbol Substitution Test | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on The Digit Symbol Substitution Test
  Wechsler, D., (2008). Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio, TX: NCS Pearson.
The Hopkins Verbal Learning Test-Revised | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on The Hopkins Verbal Learning Test-Revised
  Benedict, R. H. B., Schretlen, D., Groninger, L., & Brandt, J. (1998). The Hopkins verbal learning test-revised: Normative data and analysis of interform and test-retest reliability. Clinical Neuropsychologist, 12, 43-55.
The Rey-Osterrieth Complex Figure Test | Treatment change from Baseline to Immediate post, and 8 weeks post treatment completion.
  Evaluation of treatment differences in change on The Rey-Osterrieth Complex Figure Test
  Rey, A. (1941). L'examen psychologique dans les cas d'encéphalopathie traumatique. (Les problems.). [The psychological examination in cases of traumatic encepholopathy. Problems.]. Archives de Psychologie, 28, 215- 285.

CONTACTS AND LOCATIONS:
Overall Officials: John Hart, MD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas at Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Dugas CS, Chiang HS, Devora P, Lucas-Mendoza K, Abasi C, Adhikari A, Nguyen T, Frolov A, Kelley BJ, LoBue C, Mudar RA, Hart J Jr. High-definition brain stimulation targeting separate regions leads to differential word retrieval outcomes in patients with primary progressive aphasia: a pilot study. Front Neurol. 2025 Sep 17;16:1630103. doi: 10.3389/fneur.2025.1630103. eCollection 2025. PMID 41041680